CLINICAL TRIAL: NCT06903312
Title: Clinical and Humoral Impact of Primary Tumor Ablation in Metastatic Renal Cell Carcinoma Treated With Immunotherapy. The ITALIC-RCC Randomized Study.
Brief Title: Primary Tumor Ablation and Outcome in Metastatic Renal Cell Carcinoma Treated With Immunotherapy Combinations.
Acronym: ITALIC-RCC
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: AIRC (Italian Association for Cancer Research) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7056
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Renal Cell Cancer; Kidney Neoplasm; Immunotherapy; Kidney Cancer; Surgery Programmed; Radiotherapy
Keywords: renal cancer; primary tumor; cytoreductive nephrectomy; immunothreapy; radiotherapy
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — Radiotherapy; Nutrition Therapy; Standard of Care

STUDY DESIGN:
Intervention Model Description: Patients will be valuated for local therapy (ie: surgery or radiotherapy) while they are receiving immunotherapy-based therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Radiotherapy (Experimental): Patients with tumors up to 4 cm can receive RT single shot of 25 Gy (or with multiple fractions with equivalent biological dose).
  Interventions: Radiation: Radiotherapy + medical treatment
- Deferred Cytoreductive Nephrectomy (Experimental): Patients randomized to Deferred Cytoreductive Nephrectomy can be treated with one among radical nephrectomy; partial nephrectomy or lumpectomy.
  Interventions: Procedure: Deferred Cytoreductive Nephrectomy + medical treatment
- Control (Active Comparator): patients in the control arm continue to receive immuno-based medical treatment for mRCC.
  Interventions: Drug: Medical therapy

INTERVENTIONS:
Procedure: Deferred Cytoreductive Nephrectomy + medical treatment — Patients randomized to Deferred Cytoreductive Nephrectomy can be treated with one among radical nephrectomy; partial nephrectomy or lumpectomy. Patients will continue to receive the ongoing medical treatment before the randomization.
  Arms: Deferred Cytoreductive Nephrectomy
Radiation: Radiotherapy + medical treatment — Patients randomized to RT should be treated with single shot of 25 Gy (or with multiple fractions with equivalent biological dose). Patients will continue to receive the ongoing medical treatment before the randomization.
  Arms: Radiotherapy
Drug: Medical therapy — Medical therapy is the continuation of the immune-based combo for mRCC including one of the available options among axitinib + pembrolizumab or cabozantinib + nivolumab or lenvatinib + pembrolizumab or nivolumab alone after nivolumab + ipilimumab.
  Other Names: Standard of Care (SOC)
  Arms: Control

SUMMARY:
This is Phase IV, randomized, multi arm, multicenter, low interventional clinical trial, aiming to evaluate if treatment of primary tumor in mRCC patients with initial benefit to anti-PD1- based therapy (SOC) can improve the overall survival.

All patients eligible according to inclusion and exclusion criteria will be enrolled and randomized to different treatment options based on tumor extension of the primary kidney cancer.

Those with primary kidney cancer ≤ 4 cm will be randomized 1:1:1 to receive:

* Cytoreductive Nephrectomy + standard of care (SOC) or
* RT on primary tumor + SOC or SOC alone.

Those with primary kidney cancer > 4 cm will be randomized 1:1 to receive:

• Deferred Cytoreductive Nephrectomy + SOC or SOC alone. Patients randomized to Deferred Cytoreductive Nephrectomy can be treated with one among radical nephrectomy; partial nephrectomy or lumpectomy.

Patients randomized to RT should be treated with single shot of 25 Gy (or with multiple fractions with equivalent biological dose).

The SOC medical therapy is the continuation of the combination of medical therapy for mRCC including one of the available combination among axitinib + pembrolizumab or cabozantinib + nivolumab or lenvatinib + pembrolizumab or nivolumab alone after nivolumab + ipilimumab.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained before any study-specific procedures. Patients must be able to understand and be willing to sign a written informed consent.
2. Male or female patient ≥18 years of age.
3. Histological or cytological documentation of renal cell carcinoma with predominantly clear cell histology.
4. Evidence of primary renal cancer.
5. Measurable or not measurable metastatic disease according to Response Evaluation Criteria in Solid Tumors criteria, version 1.1 [22].
6. Eastern Cooperative Oncology Group performance status of ≤1.
7. Life expectancy of at least 9 months.
8. Under treatment with one anti-PD1 based therapy (SOC) among axitinib + pembrolizumab or cabozantinib + nivolumab or lenvatinib + pembrolizumab or nivolumab alone after nivolumab + ipilimumab for at least 24 but not more than 52 weeks at the time of the signed informed consent and without evidence of progressive disease based on RECIST criteria v 1.1 [21].
9. Eligible to continue the combination of therapies for mRCC (or nivolumab alone in case of nivolumab + ipilimumab).
10. Women of childbearing potential and men must agree to use adequate contraception since signing of the informed consent form until at least 3 months after the last study drug administration. The investigator or a designated associate is requested to advise the subject how to achieve an adequate birth control. Adequate contraception is defined in the study as any medically recommend method (or combination of methods) as per standard of care.
11. Adequate bone-marrow, liver, and renal function as assessed by the following laboratory requirements conducted within 7 days of starting to study treatment:

    1. Creatinine value <2.5 mg/dl and creatinine clearance > 30 ml/min evaluated by the Cockcroft-Gault Formula.
    2. Total bilirubin ≤1∙5 × the upper limit of normal (ULN);
    3. Alanine aminotransferase and aspartate aminotransferase ≤2 × ULN (≤5 × ULN for patients with liver involvement of their cancer);
    4. International normalized ratio (INR) and partial thromboplastin time (PTT) ≤1∙5 × ULN. Subjects who are therapeutically treated with an agent such as warfarin or heparin will be allowed to participate if no prior evidence of an underlying abnormality in coagulation parameters exists. Close monitoring of at least weekly evaluations will be performed until INR and PTT are stable based on a pre-dose measurement as defined by the local standard of care;
    5. Platelet count ≥100 000/mm3, hemoglobin >9 g/dl, absolute neutrophil count >1,500/mm3;
    6. Alkaline phosphatase limit ≤2∙5 × ULN (≤5 × ULN for patients with liver involvement of their cancer).

Exclusion Criteria:

1. More than one treatment for metastatic or locally advanced renal cell carcinoma.
2. Solitary kidney
3. Any contraindication to surgery or radiotherapy on primary renal tumor.
4. Discontinuation (definitive) of one of the therapies for mRCC due to toxicity (previous discontinuation of ipilimumab in the ipilimumab + nivolumab combo is allowed).
5. Concurrent or previous cancer within 3 years before enrolment EXCEPT curatively treated cervical cancer in situ, non-melanoma skin cancer and pT2 prostate cancer with PSA<0.01 or non-muscle invasive bladder cancer.
6. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days before the signed informed consent.
7. Pregnancy or breast-feeding. Women of childbearing potential must have a pregnancy test performed a maximum of 7 days before surgery or radiotherapy on primary tumor, and a negative result must be documented before start of treatment.
8. Any cardiological condition among:

   1. Congestive heart failure of New York Heart Association class 3 or worse.
   2. Unstable angina (angina symptoms at rest), new-onset angina (begun within the last 3 months). Myocardial infarction less than 6 months before start of study drug.
   3. Cardiac arrhythmias requiring anti-arrhythmic therapy (beta-blockers or digoxin are permitted).
   4. Uncontrolled hypertension (systolic blood pressure >150 mmHg or diastolic pressure >90 mmHg despite optimal medical management).
   5. Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), pulmonary embolism within the 4 months before start of study.
9. Ongoing infection higher than National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 6.0 grade 2.
10. Known history of human immunodeficiency (HIV) virus infection or known history of chronic hepatitis B or C.
11. Any autoimmune reaction or toxicity that contraindicates the use of anti-PD1 therapy.
12. Seizure disorder requiring medication.
13. Symptomatic metastatic brain or meningeal tumors unless the patient is >2 months from definitive therapy, has a negative imaging study within 4 weeks of study entry and is clinically stable with respect to the tumor at the time of study entry. Also, the patient must not be undergoing acute steroid therapy or tapering (chronic steroid therapy is acceptable provided that the dose is stable for 1 month before and after screening radiographic studies).
14. History of organ allograft.
15. Evidence or history of bleeding diathesis. Any hemorrhage or bleeding event of CTCAE grade 3 or higher within 4 weeks of start of study medication.
16. Non-healing wound, ulcer, or bone fracture.
17. Renal failure requiring hemodialysis or peritoneal dialysis.
18. Any illness or medical conditions that are unstable or could jeopardize the safety of the patient and his or her compliance in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 409 (Estimated)
Dates: Start 2025-06-15 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
30-months Overall Survival for surgery vs. control | 30 months
  The primary endpoint of the study is to assess the difference in 30-months overall survival (OS) between patients who receive or not the deferred citoreductive nephrectomy (CN) while on therapy with SOC for mRCC.

SECONDARY OUTCOMES:
Median overall survival for surgery vs. control | 30 months
  To assess the difference in overall survival (OS) between patients who receive or not the deferred citoreductive nephrectomy (CN) while on therapy with SOC for mRCC from the beginning of the anti-PD1-based therapy.
Median Progression Free Survival for surgery vs. control | 30 months
  To assess the difference in progression-free survival (PFS) between patients who receive or not the deferred citoreductive nephrectomy (CN) while on therapy with SOC for mRCC.
Median Overall Survival for radiotherapy vs. control | 30 months
  To assess the difference in overall survival (OS) between patients who receive or not the radiotherapy on primary tumor while on therapy with SOC for mRCC among those with primary tumor up to 4 cm at randomization.
Median Progression Free Survival for radiotherapy vs. control | 30 months
  To assess the difference in progression-free survival (PFS) between patients who receive or not the radiotherapy on primary tumor while on therapy with SOC for mRCC among those with primary tumor up to 4 cm at randomization.
Incidence of adverse events | 30 months
  To evaluate the safety of the CN and RT on primary tumor among patients receiving SOC for mRCC. Adverse events will be graded according to NCI CTCAE version 5.0.
Difference in EQ-5D-5L quality of life test | Baseline and 8 weeks after surgery or radiotherapy.
  To evaluate the quality of life before and after 8 weeks from the surgery or radiotherapy on primary tumor among patients receiving SOC for mRCC evaluated by the questionnaires EQ-5D-5L.
Difference in FKSI-19 quality of life test | Baseline and 8 weeks after surgery or radiotherapy.
  To evaluate the quality of life before and after 8 weeks from the surgery or radiotherapy on primary tumor among patients receiving SOC for mRCC evaluated by the questionnaires FKSI-19.
Incidence in of surgical complications. | 8 weeks after surgery
  To evaluate the incidence of surgical complications by the Clavien- Dindo classification.

OTHER OUTCOMES:
Difference in the proteomic profile | Before and 8 weeks after surgery or radiotherapy.
  The study aims also to describe the change of proteome after surgery or radiotherapy on primary tumor compared to the baseline and to evaluate if specific proteome profiles at baseline are related to different outcomes. A blood tumor sample will be performed at the time of randomization for all patients and after eight weeks from CN or the end of RT to assess the proteomic profile.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Iacovelli, M.D.; Ph.D., Principal Investigator — Catholic University of Rome, Italy
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No
Not planned at this time.